CLINICAL TRIAL: NCT02060760
Title: Use of Abbott High Sensitivity Troponin I Assay In Acute Coronary Syndromes
Acronym: UTROPIA
Status: Completed | Type: Observational
Sponsor: Hennepin Healthcare Research Institute (Other)
Collaborators: Abbott Diagnostics Division (Industry); Hennepin County Medical Center, Minneapolis (Other)
Responsible Party: Principal Investigator, Fred Apple, PhD, Hennepin Healthcare Research Institute
Other Study IDs: HSR 13-3690
Record Dates: First submitted 2014-02-05; First posted 2014-02-12 (Estimated); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction; Troponin
Keywords: Prospective cohort study; Diagnostic accuracy; High sensitivity versus contemporary troponin I assay; Gender; Renal Function
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 180 Days
Biospecimen Retention: Samples Without DNA — Excess blood is biobanked as EDTA-plasma and heparin samples after being used for the clinical cTnI assay according to IRB approval HSR # 07-2854
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- UTROPIA study cohort: At least two cTnI data points available (including baseline) with blood samples available for hs-cTnI testing. No intervention.

SUMMARY:
Hypothesis: High sensitivity cTnI assays will have improved diagnostic accuracy for type 1 MI compared to contemporary cTnI assays.

The primary objective of the study is to determine the performance of a high sensitivity cardiac troponin I (hs-cTnI) assay compared to a contemporary cTnI assay for the diagnostic accuracy of type 1 acute myocardial infarction (AMI).

The diagnostic performance of Abbott's hs-cTnI assay will be evaluated. Investigators will assess the assay's ability to diagnose AMI earlier and to rule out AMI earlier. The sensitivity, specificity, positive predictive value and negative predictive value of the hs-cTnI assay will be evaluated with both a universal cut off as well as with gender and potentially age derived 99th percentile upper reference limits (URL).

Investigators will evaluate delta hs-cTnI values (pre-specified absolute concentration and percent changes over time) for their ability to contribute to the negative predictive value and hence potentially lead to an earlier rule out of AMI (improved specificity). Additionally, investigators will assess delta changes of the hs-cTnI assay for their potential contribution to the clinical differentiation of type 1 and type 2 (supply demand mismatch) MIs.

Lastly, investigators will compare the diagnosis of AMI based on the currently used contemporary assay to the hs-assay, to assess both the incidence of AMI as well as for the time to diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Two or more cTnI values ordered for any clinical indication with specimen available for hs cTnI assay
* 18 years of age or older
* EKG done on admission / presentation
* Agree to research disclosure

Exclusion Criteria:

* Admission through any venue other an emergency department
* Repeat admission for the same patient, only primary admission will be assessed
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting to Hennepin County Medical Center through the emergency department within the defined study period will be considered for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 1927 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Acute Myocardial Infarction | Up to 6 months after last enrollment
  Adjudicated diagnosis of acute myocardial infarction (AMI) to systematize the potentially earlier (0,3,6h) detection of AMI using the Abbott hs cTnI assay.

SECONDARY OUTCOMES:
In- hospital mortality | Up to 6 months after last enrollment
180 day mortality | Up to 6 months after last enrollment
Repeat Cardiac hospitalization | Up to 6 months after last enrollment
Time to repeat cardiac hospitalization | Up to 6 months after last enrollment
ACS Diagnosis | Up to 6 months after last enrollment
Repeat revascularization (bypass surgery versus percutaneous revascularization) | Up to 6 months after last enrollment
Emergency encounter for chest pain | Up to 6 months after last enrollment
New diagnosis of Congestive Heart Failure | Up to 6 months after last enrollment

OTHER OUTCOMES:
Resource utilization | Up to 6 months after last enrollment
  Resource utilization rates including medications (sorted by class), cardiac evaluation procedures(e.g. echocardiogram, angiography, interventions) and speciality consultations will be assessed.
Type 2 AMI Physiologic Assessment | Up to 6 months after last enrollment
  Expert adjudication of the cause of decreased oxygen supply or increased myocardial oxygen demand resulting in positive cTnI measured by both hs-cTnI and contemporary cTnI assays based on pre-specified subtypes, including:
  * Decreased Supply
  * Increased Demand
  * Multifactorial of Indeterminate myocardial injury
Troponin in Angiography | Up to 6 months after last enrollment
  cTnI concentration changes will be analyzed among patients who underwent coronary angiography

CONTACTS AND LOCATIONS:
Overall Officials: Fred Apple, PhD, Principal Investigator — Minneapolis Medical Research Foundation and Hennepin County Medical Center
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Neumann JT, Twerenbold R, Ojeda F, Aldous SJ, Allen BR, Apple FS, Babel H, Christenson RH, Cullen L, Di Carluccio E, Doudesis D, Ekelund U, Giannitsis E, Greenslade J, Inoue K, Jernberg T, Kavsak P, Keller T, Lee KK, Lindahl B, Lorenz T, Mahler SA, Mills NL, Mokhtari A, Parsonage W, Pickering JW, Pemberton CJ, Reich C, Richards AM, Sandoval Y, Than MP, Toprak B, Troughton RW, Worster A, Zeller T, Ziegler A, Blankenberg S; ARTEMIS study group. Personalized diagnosis in suspected myocardial infarction. Clin Res Cardiol. 2023 Sep;112(9):1288-1301. doi: 10.1007/s00392-023-02206-3. Epub 2023 May 2. PMID 37131096
- [Derived] Sandoval Y, Smith SW, Sexter A, Gunsolus IL, Schulz K, Apple FS. Clinical Features and Outcomes of Emergency Department Patients With High-Sensitivity Cardiac Troponin I Concentrations Within Sex-Specific Reference Intervals. Circulation. 2019 Apr 2;139(14):1753-1755. doi: 10.1161/CIRCULATIONAHA.118.038284. No abstract available. PMID 30933618
- [Derived] Sandoval Y, Gunsolus IL, Smith SW, Sexter A, Thordsen SE, Carlson MD, Johnson BK, Bruen CA, Dodd KW, Driver BE, Jacoby K, Love SA, Moore JC, Scott NL, Schulz K, Apple FS. Appropriateness of Cardiac Troponin Testing: Insights from the Use of TROPonin In Acute coronary syndromes (UTROPIA) Study. Am J Med. 2019 Jul;132(7):869-874. doi: 10.1016/j.amjmed.2019.01.043. Epub 2019 Mar 5. PMID 30849383
- [Derived] Cediel G, Sandoval Y, Sexter A, Carrasquer A, Gonzalez-Del-Hoyo M, Bonet G, Boque C, Schulz K, Smith SW, Bayes-Genis A, Apple FS, Bardaji A. Risk Estimation in Type 2 Myocardial Infarction and Myocardial Injury: The TARRACO Risk Score. Am J Med. 2019 Feb;132(2):217-226. doi: 10.1016/j.amjmed.2018.10.022. Epub 2018 Nov 9. PMID 30419227
- [Derived] Gunsolus I, Sandoval Y, Smith SW, Sexter A, Schulz K, Herzog CA, Apple FS. Renal Dysfunction Influences the Diagnostic and Prognostic Performance of High-Sensitivity Cardiac Troponin I. J Am Soc Nephrol. 2018 Feb;29(2):636-643. doi: 10.1681/ASN.2017030341. Epub 2017 Oct 27. PMID 29079658
- [Derived] Sandoval Y, Smith SW, Thordsen SE, Bruen CA, Carlson MD, Dodd KW, Driver BE, Jacoby K, Johnson BK, Love SA, Moore JC, Sexter A, Schulz K, Scott NL, Nicholson J, Apple FS. Diagnostic Performance of High Sensitivity Compared with Contemporary Cardiac Troponin I for the Diagnosis of Acute Myocardial Infarction. Clin Chem. 2017 Oct;63(10):1594-1604. doi: 10.1373/clinchem.2017.272930. Epub 2017 Jul 12. PMID 28701316
- [Derived] Sandoval Y, Smith SW, Shah AS, Anand A, Chapman AR, Love SA, Schulz K, Cao J, Mills NL, Apple FS. Rapid Rule-Out of Acute Myocardial Injury Using a Single High-Sensitivity Cardiac Troponin I Measurement. Clin Chem. 2017 Jan;63(1):369-376. doi: 10.1373/clinchem.2016.264523. Epub 2016 Nov 3. PMID 27811203